CLINICAL TRIAL: NCT03394261
Title: Pilot Test of Patient Decision Aid for Medication-Assisted Treatment for Opioid Use Disorder
Brief Title: Pilot Test of Patient Decision Aid for Opioid Use Disorder
Acronym: PtDA-MAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OPIOD1
Record Dates: First submitted 2018-01-03; First posted 2018-01-09 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Opioid Use Disorder
Keywords: Opioid Use Disorder (OUD); Medication Assisted Therapy (MAT); Patient Decision Aid
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: The Patient Decision Aid for Medication Assisted Therapy (PtDA-MAT) will be pilot-tested by patients and clinicians during actual visits with OUD patients to assess its acceptability and feasibility. We will track patients receiving PtDAT-MAT using their clinical and administration data over a 3-month period and compare outcomes to those of treatment admissions during the 3 months prior to the pilot testing to assess preliminary outcomes associated with PtDAT-MAT.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Decision Aid (Experimental): Patients in this arm will receive Patient Decision Aid for Medication Assisted Treatment for opioid use disorder.
  Interventions: Behavioral: Patient Decision Aid
- Record-only control group (No Intervention): Treatment records of patients receiving treatment in the same clinic in the prior 3 months will be abstracted for comparison purposes.

INTERVENTIONS:
Behavioral: Patient Decision Aid — PtDA-MAT will provide information on MAT treatment options and pros and cons of each treatment option, and will assess patients' preferred options.
  Arms: Patient Decision Aid

SUMMARY:
The aims of the current study phase (R21) are: Aim 1. Develop a patient decision aid (PtDA-MAT) by incorporating best available scientific evidence on MAT as well as feedback from patients and clinical providers related to clinical priorities, perceived utility, and acceptability; Aim 2. Conduct pilot testing of the PtDA-MAT in an iterative process guided by an expert panel and involving key stakeholders (e.g., patients, physicians, policymakers) and field-testing.

DETAILED DESCRIPTION:
In response to RFA-DA-18-005 (Expanding Medication Assisted Treatment for Opioid Use Disorders in the Context of the SAMHSA Opioid STR Grants, R21/R33), this project will develop and test a patient decision support tool called Patient Decision Aid for Medication-Assisted Treatment (PtDA-MAT) for use in the CA H&SS. The PtDA-MAT is designed to (1) improve patient knowledge and involvement and to subsequently improve treatment adherence and outcomes and (2) to support clinicians in informing and communicating with their patients with OUD along a continuum of care. The project will conduct 1 year of R21 to develop and pilot-test the PtDA-MAT to facilitate shared decision making in CA H&SS, followed by 3 years of R33 to assess the effectiveness of the PtDA-MAT in a randomized controlled trial.

The aims of the current study phase (R21) are: Aim 1. Develop a patient decision aid (PtDA-MAT) by incorporating best available scientific evidence on MAT as well as feedback from patients and clinical providers related to clinical priorities, perceived utility, and acceptability; Aim 2. Conduct pilot testing of the PtDA-MAT in an iterative process guided by an expert panel and involving key stakeholders (e.g., patients, physicians, policymakers) and field-testing.

ELIGIBILITY:
Inclusion Criteria:

* Opioid Use Disorder diagnosis and agreement to follow study procedures (including permission to share medical records and other administrative records)

Exclusion Criteria:

* Significant or unstable medical or psychiatric illness that may interfere with study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-06-14 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2018-12-21 (Actual)

PRIMARY OUTCOMES:
Treatment Retention | 3 months
  Treatment retention will be defined as number of days from initial treatment admission to either MAT discontinuation or most recent clinic visit followed by 2 months gap in treatment

SECONDARY OUTCOMES:
Drug screening results | 3 month
  Primarily opioid-negative urine testing (as collected by clinics as part of routine care) and other substance use per self-report (e.g., cannabis, benzodiazepines, cocaine, amphetamines)
Treatment Adherence | 3 month
  Treatment Adherence defined as proportion of clinic visits attended

CONTACTS AND LOCATIONS:
Overall Officials: Yih-Ing Hser, Ph.D., Principal Investigator — University of California, Los Angeles; Larissa Mooney, M.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- Tarzana Treatment Centers, Inc., Tarzana, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mooney LJ, Valdez J, Cousins SJ, Yoo C, Zhu Y, Hser YI. Patient decision aid for medication treatment for opioid use disorder (PtDA-MOUD): Rationale, methodology, and preliminary results. J Subst Abuse Treat. 2020 Jan;108:115-122. doi: 10.1016/j.jsat.2019.08.006. Epub 2019 Oct 24. PMID 31668516